CLINICAL TRIAL: NCT00872079
Title: Personalized Warfarin Dosing Using Genomics and Computational Intelligence
Brief Title: Personalized Warfarin Dosing by Genomics and Computational Intelligence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CAMM-04-07S
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Venous Thrombosis; Atrial Fibrillation; Myocardial Infarction
Keywords: warfarin; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Venous Thrombosis; Atrial Fibrillation; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genomics (Active Comparator): Aim 1: Collect historical data on warfarin dosing in subjects at the VA. Aim 2: Collect genotype information on up to 300 subjects receiving warfarin anticoagulation.
  Aim 3: Develop a computer model incorporating the information from Aim 1 and 2. Aim 4: Conduct randomized clinical trial.
  Interventions: Device: Genomics

INTERVENTIONS:
Device: Genomics — Model predictive control is a computer based algorithm that can be applied to drug dosing. This computer tool uses a model of how a patient will respond to a drug dose based on demographic and historical dosing information to predict a new drug response. A drug dose controller applies all possible doses to the response model and selects the one dose that best meets the stated goals of the drug therapy. In the case of warfarin, we will calculate an international normalized ratio (INR) value within a specific target range.

SUMMARY:
This study will create a computer program that can be used to help dose a drug called warfarin for the prevention of blood clotting. The study will collected specific information about those patients receiving this drug and use that information to create a computer program that will predict the effects of the drug. With this prediction program in place, the investigators can perform a series of "what if I gave this amount of drug" simulations to determine the best dose of drug for that patient. Once the computer programs are developed, the investigators will test the program in patients that actually need this drug. They will also include genetic information into the prediction since it has been shown that this information can affect how well the drug works. Patients will have this genetic information determined during this study.

DETAILED DESCRIPTION:
The objective of this project is to develop new techniques to incorporate genomic data into pharmacodynamic models to improve the dosing of chronically administered drugs. Specifically, the investigators look to improve warfarin therapy by decreasing the variability in the effect of this drug using information about the subjects genotype and computational intelligence. The investigators propose to achieve our objectives using a prospective, randomized, controlled clinical trial of a computer program that they will develop from both historical and prospective data. This computer program will be tested against a control group using standard warfarin dosing, and a group using standard dosing plus subject genotype. Warfarin dose and response data will be obtained from patients seen in the Louisville VA anticoagulation clinic. Following informed consent, subject genotype for cytochrome P450 allele 2C9 (2C9) and vitamin K epoxide reductase complex subunit 1 (VKORC1) will be determined. Other data routinely obtained to aid in warfarin dosing will also be recorded. Using this information, the investigators will develop many different models for warfarin dosing using incrementally more information. Each of these models will be tested using computer simulation until they have obtained the best model. This model will be used in a pilot study to test performance in real time. The results of the pilot study will then be used to power a final clinical trial of standard dosing, standard dosing and genetic information, computer dosing, and computer dosing plus genetic information.

The specific aims of this research are:

1. Determine the structure and the type of neural network model for predictions from historically obtained data. (Computer Model)
2. Prospectively develop an individualized neural network and nonlinear mixed effect modelling (NONMEM) model capable of predicting erythropoietin dosing for chronic in-center hemodialysis patients using adaptive techniques.
3. Develop computer programs based on neural computing that can be used in a clinical setting. (Computer Model)
4. Determine the utility of the computer programs prospectively in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Warfarin therapy
* Attend anticoagulation clinic
* Warfarin therapy for 6 months

Exclusion Criteria:

* History of non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Brier, PhD, Principal Investigator — VA Medical Center, Louisville
Locations (1):
- VA Medical Center, Louisville, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not enrolled into the randomized clinical trial for Aim 4 due to lack of funding.
Groups:
- Genomics: Model Predictive Control: Model predictive control is a computer based algorithm that can be applied to drug dosing. This computer tool uses a model of how a patient will respond to a drug dose based on demographic and historical dosing information to predict a new drug response. A drug dose controller applies all possible doses to the response model and selects the one dose that best meets the stated goals of the drug therapy. In the case of warfarin, we will calculate an INR value within a specific target range.
Period: Overall Study
Arm/Group | Genomics
Started | 175
Completed | 175
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Genomics: The specific aims of this research are:
  1. Determine the structure and the type of neural network model for predictions from historically obtained data. (Computer Model)
  2. Prospectively develop an individualized neural network and NONMEM model capable of predicting erythropoietin dosing for chronic in-center hemodialysis patients using adaptive techniques.
  3. Develop computer programs based on neural computing that can be used in a clinical setting. (Computer Model)
  4. Determine the utility of the computer programs prospectively in the clinical setting.
Arm/Group | Genomics
Number analyzed (Participants) | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 125
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 165
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 17
  White | 157
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Genomics
Description: During Aim 2, Determined Patient Genotypes: CYP2C9 and VKORC1.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Genomics: Model Predictive Control: Model predictive control is a computer based algorithm that can be applied to drug dosing. This computer tool uses a model of how a patient will respond to a drug dose based on demographic and historical dosing information to predict a new drug response. A drug dose controller applies all possible doses to the response model and selects the one dose that best meets the stated goals of the drug therapy. In the case of warfarin, we will calculate an INR value within a specific target range.
  There are 4 Aims in this study.
  1. To collect historical data on warfarin dosing in subjects.
  2. To collect genotype information on up to 300 subjects receiving warfarin anticoagulation.
  3. to develop a computer model incorporating the information from aim 1 and aim 2.
  4. To conduct a randomized clinical trial.
Arm/Group | Genomics
Number analyzed (Participants) | 175
participants
  CYP2C9: *1/*1 | 112
  CYP2C9: *1/*2 | 23
  CYP2C9: *1/*3 | 19
  CYP2C9: *2/*2 | 3
  CYP2C9: *2/*3 | 3
  CYP2C9: *3/*3 | 2
  CYP2C9: Not Determined | 13
  VKORC1: AA | 23
  VKORCI:GA | 72
  VKORCI:GG | 67
  VKORCI: Not Determined | 13

ADVERSE EVENTS:
Arm/Group | Genomics
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No